CLINICAL TRIAL: NCT05546749
Title: Virtual Reality Treatment in a Methadone Maintenance Treatment Program for Chronic Pain and Opioid Use Disorder
Brief Title: Virtual Reality for Chronic Pain and Opioid Use Disorder Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-14257; 1R01DA060796-01 (NIH)
Record Dates: First submitted 2022-09-13; First posted 2022-09-21 (Actual); Results first posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Chronic Pain; Opioid Use Disorder
MeSH Terms: conditions — Chronic Pain; Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- RelieVRx (Active Comparator): RelieVRx was designed for at-home use and comes with a sequence of daily immersive experiences. Participants in the intervention group will complete 20-30 minute VR sessions twice per week over the course of 6 weeks.
  Interventions: Device: RelieVRx
- Sham Virtual Reality (Sham Comparator): The sham virtual reality (VR) device is also by RelieVRx. However, it lacks the immersive nature of the interventional VR. Control participants will complete 20-30 minute VR sessions twice per week over the course of 6 weeks.
  Interventions: Device: Sham VR

INTERVENTIONS:
Device: RelieVRx — The virtual reality device that will be piloted is called RelieVRx, which incorporates evidence-based principles of cognitive behavioral therapy, mindfulness, and pain neuroscience education into an immersive and enhanced biofeedback experience. RelieVRx includes breathing training and relaxation response exercises that activate the parasympathetic nervous system. RelieVRx was designed for at-home use and comes with a sequence of daily immersive experiences.
  Arms: RelieVRx
Device: Sham VR — The sham VR control is a non-immersive set of 56 daily virtual experiences, tuned to the length of the RelieVRx.
  Arms: Sham Virtual Reality

SUMMARY:
This is a pilot feasibility study of a virtual reality device for patients with co-morbid chronic pain and opioid use disorder.

DETAILED DESCRIPTION:
The investigators will conduct a study of patients with co-morbid chronic pain and opioid use disorder enrolled in a methadone maintenance treatment program (MMTP) to pilot device feasibility and measure changes in pain intensity and opioid craving. All patients will be randomized to one of each of the following arms: 1) RelieVRx (intervention group) or 2) Non-immersive sham VR (control group).

The intervention being piloted is the RelieVRx - AppliedVR, Los Angeles, California - VR hardware and software. RelieVRx incorporates evidence-based principles of cognitive behavioral therapy, mindfulness, and pain neuroscience education into an immersive and enhanced biofeedback experience. RelieVRx includes breathing training and relaxation response exercises that activate the parasympathetic nervous system. RelieVRx was designed for at-home use and comes with a sequence of daily immersive experiences.

RelieVRx is typically delivered in a 56-day program through daily virtual experiences, with each experience lasting between 2 and 16 minutes. In this pilot study, the investigators will conduct virtual experiences twice weekly at the MMTP. Over 6 weeks, participants in both groups will participate in 20-30 minute VR sessions twice per week. Each session will last about 20-30 minutes and go through 1-5 virtual experiences. The sham VR control is a non-immersive set of 56 daily virtual experiences, tuned to the length of the RelieVRx. Control participants will similarly experience 1-5 virtual experiences in each 20-30 session.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old
2. English proficiency
3. receiving methadone treatment for DSM-5 (Diagnostic and Statistical Manual of Mental Disorders, 5th Edition) confirmed Opioid Use Disorder (OUD) in the Montefiore network for at least 12 weeks, with no dose change in 14 days to ensure treatment stability
4. chronic pain of at least moderate pain severity (score ≥4 on the Pain, Enjoyment of Life, and General Activity (PEG) scale)
5. willingness to participate in all study components
6. ability to provide informed consent, assessed using consent teach-back

Exclusion Criteria:

1. conditions that could make participation in VR hazardous or cause adverse effects (current or prior diagnosis of epilepsy, seizure disorder, dementia, or migraines, any medical condition predisposing to nausea or dizziness, hypersensitivity to flashing light or motion)
2. conditions that could prevent proper use of the VR headset (stereoscopic vision or severe hearing impairment, or injury to eyes, face, or neck that prevents use of the VR headset)
3. acute exacerbation of psychiatric conditions that preclude the ability to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-02-08 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2023-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hector Perez, MD, MS, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Melrose Clinic, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RelieVRx | Sham Virtual Reality
Started | 10 | 8
Completed | 8 | 6
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RelieVRx | Sham Virtual Reality | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (5.3) | 60.3 (8.0) | 59.8 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 5 | 2 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, non-Hispanic | 0 | 1 | 1
  Black, non Hispanic | 4 | 3 | 7
  Hispanic, any race | 6 | 4 | 10
Region of Enrollment [Number; unit: participants]
  United States | 10 | 8 | 18
Education [Count of Participants; unit: Participants] — The number of participants who did not complete High School (HS), completed their General Educational Development (GED) or equivalent, received their HS diploma, or completed 1 or more years of college/university were summarized by study arm.
  Participants
    Did not complete High School (HS) | 3 | 3 | 6
    Completed GED or equivalent | 3 | 0 | 3
    Received HS diploma | 2 | 4 | 6
    Completed 1 or more years of college/university | 2 | 1 | 3
Pain impact (PEG score) [Mean (Standard Deviation); unit: score on a scale] — Pain, Enjoyment of Life, and General Activity (PEG) scale scores were obtained at baseline. The PEG score is a 3-item pain assessment tool that measures the impact of pain intensity and interference on a participant's daily life. The PEG score is calculated by averaging the responses to three questions each on a scale of 0-10. Higher average (mean) scores are associated with increased impact of pain on a participant's life. Scores were summarized by study arm using basic descriptive statistics.
  score on a scale | 7.67 (1.67) | 6.71 (1.86) | 7.24 (1.78)

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Intensity
Description: Change in Pain Intensity from baseline was assessed using the single items Patient-Reported Outcomes Measurement Information System (PROMIS) pain intensity scale. Patients were asked to assess their average pain over the past 7 days on an 11-point Likert scale ranging from 0-10 where 0 = no pain and 10 = worst pain imaginable. Positive mean scores were associated with increased pain intensity from baseline and negative mean scores were associated with decreased pain intensity from baseline. Scores were summarized by study arm using basic descriptive statistics.
Time Frame: From baseline to 6 weeks
Population: 8 participants in the RelieVRx arm and 6 participants in the Sham Virtual Reality arm completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RelieVRx | Sham Virtual Reality
Number analyzed (Participants) | 8 | 6
score on a scale | -1.38 (1.69) | 0.33 (2.66)
Statistical Analysis 1: Comparison: RelieVRx vs Sham Virtual Reality; A mixed effects model was performed to predict pain intensity by arm at weeks 3 and 6, controlling for baseline pain intensity score; Test type: Superiority; p = 0.17, Mixed Models Analysis; Mean Difference (Final Values) = -1.28, 95% CI 2-sided [-3.1 to 0.54], Standard Error of Mean .93

2. Primary Outcome: Change in Opioid Craving
Description: Change in Opioid Craving was assessed using the Opioid Medication Craving Visual Analog Scale. This 3-item scale asked participants to rate how strong their desire to use opioids was during the previous 24 hours; the likelihood that they would use opioids if placed in the environment in which they had previously used drugs/alcohol; and how strong their urges for opioids are when something in their environment reminds them of it. Responses were marked on visual scale ranging from 0-100 where "0" signified 'No Desire or Likelihood of Use' and "100" signified 'Strong Desire or Likelihood of use. Positive mean scores were associated with increased opioid craving from baseline and negative mean scores were associated with decreased opioid craving from baseline. Scores were summarized by study arm using basic descriptive statistics.
Time Frame: From baseline to 6 weeks
Population: 8 participants in the RelieVRx arm and 6 participants in the Sham Virtual Reality arm completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RelieVRx | Sham Virtual Reality
Number analyzed (Participants) | 8 | 6
score on a scale | -2.86 (30.9) | 9.17 (17.44)
Statistical Analysis 1: Comparison: RelieVRx vs Sham Virtual Reality; A mixed effects model was used to predict opioid craving score by arm at weeks 3 and 6, controlling for baseline opioid craving score; Test type: Superiority; p = 0.32, Mixed Models Analysis; Mean Difference (Final Values) = -13.6, 95% CI 2-sided [-40.3 to 13.1], Standard Error of Mean 13.6

3. Primary Outcome: Percentage of Participants Contacted That Are Enrolled
Description: The percentage of participants contacted who were enrolled into the study was used to assess the feasibility of the study. Results were summarized using basic descriptive statistics.
Time Frame: Baseline, up to 2 weeks
Population: All participants who were contacted enrolled into the study.
Measure: Count of Participants; unit: Participants
Arm/Group | RelieVRx | Sham Virtual Reality
Number analyzed (Participants) | 10 | 8
Participants | 10 | 8

4. Secondary Outcome: Change in Pain Interference
Description: Change in pain interference was assessed using the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference Short Form 4a scale. This form consists of 4 items which asked participants to rate the degree to which their pain interfered with a range of activities over the prior 7 days. Responses to the 4 items are summed up on a 5-point Likert scale ranging from "Not at all" = 0 to "Very much" = 4, for an overall possible scoring range of 0-16 such that higher scores are associated with greater pain interference. For purposes of reporting of this change from baseline outcome measure, positive mean scores were associated with greater pain interference relative to baseline and negative mean scores were associated with reduced pain interference relative to baseline. Scores were summarized by study arm using basic descriptive statistics.
Time Frame: From baseline to 6 weeks
Population: 3-week Pain Interference (PROMIS, Pain Interference 4a) data was not collected and, therefore, results were not available to be reported. 8 participants in the RelieVRx arm and 6 participants in the Sham Virtual Reality arm completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RelieVRx | Sham Virtual Reality
Number analyzed (Participants) | 8 | 6
score on a scale | -2.25 (8.43) | 1.67 (5.20)

5. Secondary Outcome: Change in Sleep
Description: Change in sleep was assessed using the Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance Short Form 6a. This form consists of 6 items which asked participants to assess quality and attributes of their sleep patterns over the prior 7 days. Response options for the sleep quality item range from "Very poor" = 1 to "Very good = 5" and from "Not at all" = 1 to "Very much" = 5 for the remaining five items. The two positively phrased items are reverse-coded and sum scores are calculated and the raw sum score is rescaled on the PROMIS conversion table to determine a standardized T-score (overall mean of 50 and standard deviation of 10). For purposes of reporting of this change from baseline outcome measure, positive mean scores were associated with greater sleep disturbance and decreased overall sleep quality relative to baseline and negative mean scores were associated with decreased sleep disturbance and increased overall sleep quality relative to baseline.
Time Frame: From baseline to 6 weeks
Population: 3-week Sleep (PROMIS, Sleep Disturbance 6a) data was not collected and, therefore, results were not available to be reported. 8 participants in the RelieVRx arm and 6 participants in the Sham Virtual Reality arm completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RelieVRx | Sham Virtual Reality
Number analyzed (Participants) | 8 | 6
score on a scale | 0 (8.52) | 3 (3.90)

6. Secondary Outcome: Change in Cognitive Function
Description: Change in cognitive function was assessed using the Patient-Reported Outcomes Measurement Information System (PROMIS 29) Cognitive Function domain form. This form consists of 2 questions which asked participants to assess cognitive function over the prior 7 days. Both questions for this measure are summed up on a 5-point Likert scale ranging from "Not at all" to "Very much" = 4, for an overall possible scoring range of 0-8 such that higher scores are associated with increased overall cognitive function. For purposes of reporting of this change from baseline outcome measure, positive mean scores were associated with increased overall cognitive function from baseline and negative mean scores were associated with decreased overall cognitive function from baseline. Scores were summarized by study arm using basic descriptive statistics.
Time Frame: From baseline to 6 weeks
Population: 3-week Cognitive Function (PROMIS 29 Cognitive Function) data was not collected and, therefore, results were not available to be reported. 8 participants in the RelieVRx arm and 6 participants in the Sham Virtual Reality arm completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RelieVRx | Sham Virtual Reality
Number analyzed (Participants) | 8 | 6
score on a scale | 1.5 (3.25) | -0.67 (2.50)

7. Secondary Outcome: Change in Social Function
Description: Change in social function was assessed using the Patient-Reported Outcomes Measurement Information System (PROMIS) Social 4a Heal form. This form consists of 4 items which asked participants to assess their leisure, family, work and general social function behaviors over the prior 7 days. Responses to the 4 items are summed up on a 5-point Likert scale ranging from "Never" = 0 to "Always" = 4, for an overall possible scoring range of 0-16 such that higher scores are associated with increased inhibition in social function/participation. For purposes of reporting of this change from baseline outcome measure, positive mean scores were associated with decreased inhibition to social participation relative to baseline and negative mean scores were associated with increased inhibition to social participation relative to baseline. Scores were summarized by study arm using basic descriptive statistics.
Time Frame: From baseline to 6 weeks
Population: 3-week Social Function (PROMIS, Social 4a Heal) data was not collected and, therefore, results were not available to be reported. 8 participants in the RelieVRx arm and 6 participants in the Sham Virtual Reality arm completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RelieVRx | Sham Virtual Reality
Number analyzed (Participants) | 8 | 6
score on a scale | 2 (3.51) | 0.333 (3.44)

8. Secondary Outcome: Change in Physical Function
Description: Change in physical function was assessed using the Patient-Reported Outcomes Measurement Information System (PROMIS) Social 6b Heal form. This form consists of 6 items which asked participants to assess their physical function and ability to conduct chores, climb stairs, walk, and run errands. Responses to the 6 items are summed up on a 5-point Likert scale ranging from "Without any difficulty" (or "Not at all") = 0 to "Unable to do" (or "Cannot do") = 4, for an overall possible scoring range of 0-24 such that higher scores are associated with increased inhibition in physical function. For purposes of reporting of this change from baseline outcome measure, positive mean scores were associated with decreased inhibition in physical function relative to baseline and negative mean scores were associated with increased inhibition in physical function relative to baseline. Scores were summarized by study arm using basic descriptive statistics.
Time Frame: From baseline to 6 weeks
Population: 3-week Physical Function (PROMIS, Social 6b Heal) data was not collected and, therefore, results were not available to be reported. 8 participants in the RelieVRx arm and 6 participants in the Sham Virtual Reality arm completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RelieVRx | Sham Virtual Reality
Number analyzed (Participants) | 8 | 6
score on a scale | 1.13 (5.38) | -1.83 (3.49)

9. Secondary Outcome: Change in Depression
Description: Change in depression was assessed using the Patient-Reported Outcomes Measurement Information System (PROMIS) Depression 4a Heal form. This form consists of 4 items which asked participants to assess the frequency of depressive symptoms over the prior 7 days. Responses to the 4 items are summed up on a 5-point Likert scale ranging from "Never" = 0 to "Always" = 4, for an overall possible scoring range of 0-16 such that higher scores are associated with a greater level of depression-related symptoms. For purposes of reporting of this change from baseline outcome measure, positive mean scores were associated with greater frequency of depression-related symptoms relative to baseline and negative mean scores were associated with reduced frequency of depression-related symptoms relative to baseline. Scores were summarized by study arm using basic descriptive statistics.
Time Frame: From baseline to 6 weeks
Population: 3-week Depression (PROMIS, Depression 4a Heal) data was not collected and, therefore, results were not available to be reported. 8 participants in the RelieVRx arm and 6 participants in the Sham Virtual Reality arm completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RelieVRx | Sham Virtual Reality
Number analyzed (Participants) | 8 | 6
score on a scale | -2.38 (5.01) | -2.5 (4.46)

10. Secondary Outcome: Change in Anxiety
Description: Change in anxiety was assessed using the Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety 4a Heal form. This form consists of 4 items which asked participants to assess the frequency of onset of anxiety-related symptoms over the prior 7 days. Responses to the 4 items are summed up on a 5-point Likert scale ranging from "Never" = 0 to "Always" = 4, for an overall possible scoring range of 0-16 such that higher scores are associated with a greater level of anxiety-related symptoms. For purposes of reporting of this change from baseline outcome measure, positive mean scores were associated with greater frequency of anxiety symptoms relative to baseline and negative mean scores were associated with reduced frequency of anxiety symptoms relative to baseline. Scores were summarized by study arm using basic descriptive statistics.
Time Frame: From baseline to 6 weeks
Population: 3-week Anxiety (PROMIS, Anxiety 4a Heal) data was not collected and, therefore, results were not available to be reported. 8 participants in the RelieVRx arm and 6 participants in the Sham Virtual Reality arm completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RelieVRx | Sham Virtual Reality
Number analyzed (Participants) | 8 | 6
score on a scale | -2.88 (6.64) | -1.0 (4.34)

11. Other Pre Specified Outcome: Change in Stress
Description: Change in stress was assessed using the National Institutes of Health (NIH) Perceived Stress Scale (PSS-10) which consists of 10 items asking participants to assess the frequency of onset of stress-related symptoms over the prior month on a 5-item Likert scale ranging from 0-4. Six of the ten items are coded such that "Never" = 0 and "Very often" = 4; and four of the ten items are reverse-coded such that "Never" =4 and "Very often" = 0, for an overall scoring range of 0-40. The higher the score the worse the perceived stress. For purposes of reporting of this change from baseline outcome measure, positive mean scores were associated with greater frequency of stress relative to baseline and negative mean scores were associated with reduced frequency of stress relative to baseline. Scores were summarized by study arm using basic descriptive statistics.
Time Frame: From baseline to 6 weeks
Population: 3-week Stress (NIH Perceived Stress Scale) data was not collected and, therefore, results were not available to be reported. 8 participants in the RelieVRx arm and 6 participants in the Sham Virtual Reality arm completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RelieVRx | Sham Virtual Reality
Number analyzed (Participants) | 8 | 6
score on a scale | -4.13 (8.13) | 4.17 (15.70)
Statistical Analysis 1: Comparison: RelieVRx vs Sham Virtual Reality; We performed a mixed effects model to predict stress score at week 6 by arm, controlling for baseline stress score; Test type: Superiority; p = 0.137, Regression, Linear; Mean Difference (Final Values) = -9.7, 95% CI 2-sided [-23.1 to 3.6], Standard Error of Mean 6.1 — RelieVRx was associated with lower stress score

12. Other Pre Specified Outcome: Change in Salivary Cortisol
Description: The investigators will collect saliva the morning of each time frame and test for cortisol, which is a chronic pain inflammatory biomarker. Higher levels of salivary cortisol may indicate greater chronic pain symptoms.
Time Frame: baseline, 3 weeks, 6 weeks
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Change in Serum Cortisol
Description: The investigators will collect blood and urine samples at each time frame and test for serum cortisol, which is a chronic pain inflammatory biomarker. Higher levels of serum cortisol may indicate greater chronic pain symptoms.
Time Frame: baseline, 3 weeks, 6 weeks
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Change in Serum C-reactive Protein
Description: The investigators will collect blood samples at each time frame and test for serum c-reactive protein, which is a chronic pain inflammatory biomarker. Higher levels of serum c-reactive protein may indicate greater chronic pain symptoms.
Time Frame: baseline, 3 weeks, 6 weeks
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Change in Serum Cytokines
Description: The investigators will collect blood samples at each time frame and test for serum cytokines, which is a chronic pain inflammatory biomarker. Higher levels of serum c-reactive protein may indicate greater chronic pain symptoms.
Time Frame: baseline, 3 weeks, 6 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Approximately 6 weeks
Arm/Group | RelieVRx | Sham Virtual Reality
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8
Other Adverse Events (participants affected / at risk) | 1/10 | 0/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RelieVRx (N=10) | Sham Virtual Reality (N=8)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) — Participant vomited during blood draw during last visit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-20): https://cdn.clinicaltrials.gov/large-docs/49/NCT05546749/Prot_SAP_000.pdf